CLINICAL TRIAL: NCT07320547
Title: The Effect of a Mindfulness-Based Technology Addiction Program Applied to High School Students on Mindfulness, Internet and Smartphone Addiction
Brief Title: Mindfulness-Based Technology Addiction Program
Acronym: MBTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Collaborators: Çankırı Karatekin University (Other); Scientific and Technological Research Council of Türkiye (Unknown)
Responsible Party: Principal Investigator, Hilal ALTUNDAL DURU, Assistant professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ÇankırıKU
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Technology Addiction; Internet Addiction; Smartphone Addiction
Keywords: smartphone addiction; High school student; internet addiction; mindfulness; randomized controlled study
MeSH Terms: conditions — Technology Addiction; Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-armed (1:1), randomized controlled experimental study. This randomized controlled trial will be reported according to the CONSORT-SPI guidelines.
Who Masked: Participant
Masking Description: High school students in the experimental and control groups will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Brief Self-compassion Program will be held in a face-to-face school environment for the high school students in the experimental group. The MBTAP was carried out face-to-face in the classroom for the high school students in the intervention group. The goal of the program was to improve high school students' mindfulness levels, and decrease internet and smartphone additions' levels. This program was developed based on the concepts of mindfulness. The MBTAP was created in a certain flow based on the awekening to mindfulness (2 sessions), breath, body and mind (2 sessions), mindfulness and stress (2 sessions) and power of the compassion. There are 8 sessions lasting four weeks in the program and the frequency of sessions is 2 sessions per week and each session lasts approximately 50 minutes. The training program will be applied to 64 high school students in the experimental group.
  Interventions: Other: Mindfulness-Based Technology Addiction Program
- Control group (No Intervention): There will be no training or intervention.

INTERVENTIONS:
Other: Mindfulness-Based Technology Addiction Program — The MBTAP was carried out face-to-face in the classroom for the high school students in the intervention group. The goal of the program was to improve high school students' mindfulness levels, and decrease internet and smartphone additions' levels. This program was developed based on the concepts of mindfulness. The MBTAP was created in a certain flow based on the awekening to mindfulness (2 sessions), breath, body and mind (2 sessions), mindfulness and stress (2 sessions) and power of the compassion. There are 8 sessions lasting four weeks in the program and the frequency of sessions is 2 sessions per week and each session lasts approximately 50 minutes.
  Arms: Experimental group

SUMMARY:
In this study, between 1 September 2023-31 January 2024, who met the inclusion and exclusion criteria, a total of 128 high school students in a state high school in Çankırı.

ELIGIBILITY:
Inclusion Criteria:

* being a first-year high school student studying at state high school in a central city of Türkiye
* both student and parent agreeing to participate in the study and 3) not having communication barrier

Exclusion Criteria:

* having an illness that would prevent participation in the study
* withdrawing from the research voluntarily
* not attending at least one of the sessions
* not receiving other psychological training at the time of the research
* not receiving mindfulness-based mediation experience
* incomplete answering the instruments.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Mindful Attention Awareness Scale (MAAS) | Change from before implementation, after practice is completed (4th week)
  The MAAS consists of 15 items and is 6-point Likert type (almost always (1), most of the time (2), sometimes (3), rarely (4), very rarely (5), almost never (6)). The MAAS, which measures the general tendency to be aware of and attentive to moment-to-moment experiences in daily life, has a single-factor structure and no reverse-coded questions. High scores on the scale indicate high levels of mindfulness. The Cronbach's alpha reliability coefficient was determined to be 0.80

SECONDARY OUTCOMES:
Young's Internet Addiction Test-Short Form (YIAT-SF) | Change from before implementation, after practice is completed (4th week)
  The YIAT-SF consists of 12 items, one factor and is 5-point Likert type. Scores on the form range from 12 (lowest) to 60 (highest) and a high score on the test indicates greater levels of internet addiction. The Cronbach's alpha reliability coefficient was determined to be 0.86.
Smartphone Addiction Scale-Short Version (SAS-SF) | Change from before implementation, after practice is completed (4th week)
  The SAS-SF consists of 10 items, one factor and 6-point Likert type. Scores on the scale range from 10 (lowest) to 60 (highest) and a high score on the form indicates greater levels of smartphone addiction. The Cronbach's alpha reliability coefficient was determined to be 0.90.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No